CLINICAL TRIAL: NCT06654583
Title: Effectiveness of Developed Interactive Play Mat In Pediatric Physical Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/743
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive Play Mat (Experimental)
  Interventions: Behavioral: Interactive Play Mat
- Conventional Physical Therapy (Experimental)
  Interventions: Behavioral: Conventional Physical Therapy

INTERVENTIONS:
Behavioral: Interactive Play Mat — Use of developed interactive play mat that utilizes haptic feedback vibrations to assist children with delayed milestones in achieving Gross Motor Skills. The play mat aims to provide a therapeutic and engaging experience by incorporating visuals, sounds, and lights to encourage movement that might otherwise be challenging for these children.
  Arms: Interactive Play Mat
Behavioral: Conventional Physical Therapy — Stretching and Strengthening exercises
  Arms: Conventional Physical Therapy

SUMMARY:
The proposed study seeks to innovate by harnessing the potential of an interactive play mat, integrating haptic feedback and captivating sensory stimuli, to facilitate and expedite the motor skill development process in children with delayed milestones.

DETAILED DESCRIPTION:
This research endeavors to contribute substantively to the field of pediatric therapy by providing an engaging, effective, and accessible intervention that aligns with the specific needs of this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Delayed Milestones, 2-5 Years of age

Exclusion Criteria:

* Spina Bifida, Hydrocephalus

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Gross motor function classification system | 12 Months
  GMFCS looks at movements like sitting and walking, and it provides a a clear description of someone's current motor function, and an idea of what equipment or mobility aids a child or adult may need in the future, like crutches, a walker, or a wheelchair. GMFCS Level I Can walk indoors and outdoors and climb stairs without using their hands for support.

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Azra Naheed Medical College, Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No